CLINICAL TRIAL: NCT04079907
Title: Effects of Ketone Supplementation on Functional Outcomes in Adolescents Post-Concussion
Brief Title: Ketone Supplementation in Adolescents Post-Concussion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Eric P. Plaisance, Associate Professor of Kinesiology, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KAC2019
Record Dates: First submitted 2019-07-17; First posted 2019-09-06 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Concussion, Mild; Concussion, Severe; Concussion, Brain; Concussive Injury; Sport Injury; Sports Injuries in Children
MeSH Terms: conditions — Brain Concussion | interventions — Ketones

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into 1 of 2 groups, experimental or placebo control, and will remain in that group for the duration of the study.
Who Masked: Participant
Masking Description: Participants will not be aware if the supplement they receive is the experimental supplement or the placebo control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketone (Experimental): This arm will receive a supplement with 25g ketone ester. It is a commercially available supplement and will be provided as a standard dose.
  Interventions: Dietary Supplement: Ketone
- Placebo (Placebo Comparator): This arm will receive an isocaloric supplement.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Ketone — This intervention will take their respective supplement for 14 days, then will be followed for up to 1 year during routine clinic visits.
  Arms: Ketone
Dietary Supplement: Placebo — This intervention will take their respective supplement for 14 days, then will be followed for up to 1 year during routine clinic visits.
  Arms: Placebo

SUMMARY:
Adolescent brains undergo rapid and significant changes in structural architecture and functional organization during development. A concussive injury during this developmental period can have substantial physiological and cognitive ramifications. If not adequately managed, adolescent concussions can have profound long-term effects. The purpose of this study is to determine whether ketone supplementation after a concussion will reduce long-term consequences and improve short-term functional status and outcomes in adolescents who have suffered a concussion.

DETAILED DESCRIPTION:
In this randomized design, study participants (n=30) will take a supplement 3 times per day for 14 days and will be followed throughout completion of the concussion protocol, up to one year. The initial visit (pre-experimental visit) will serve to obtain informed consent, anthropometric information, a 24-hour dietary recall, health and lifestyle questionnaire, and circulating metabolites. Randomization will also occur at the initial visit and will be done by a computer to determine each participant's group assignment. Unless otherwise specified, follow up visits (experimental visits) will involve an identical clinical protocol as described below. The following are clinical tests that will be conducted during study visits:

Initial Visit: Participants will arrive to the Concussion Clinic in the Sports Medicine Clinic at Children's of Alabama for their routine initial visit. Participants will be provided with the study protocol, the purpose of the study, and routine and potential risks associated with the study procedures. Participants will then fill out the informed consent/assent, health and lifestyle questionnaire, and 24-hour dietary recall. As part of standard of care, height and weight will be measured using a stadiometer, body mass index (BMI) will be calculated, circulating metabolites will be collected, and resting blood pressure will be measured using a standard blood pressure cuff and a stethoscope. The SCAT5 will be conducted by a licensed healthcare professional. For research-specific purposes, body composition will be measured using BIA, C3Logix evaluation will be conducted by trained research personnel, and MRI scans will be taken. Participants will then be randomly assigned to 1 of 2 experimental groups and the appropriate supplement will be provided. Participants will also be provided with information regarding Return-to-Play progression and documents to track Return-to-Learn, supplement compliance, and GI distress.

Follow-up Visits: Participants will arrive to the Concussion Clinic in the Sports Medicine Clinic at Children's of Alabama for their routine follow up visits. Participants will fill out the 24-hour dietary recall. As part of standard of care, height and weight will be measured using a stadiometer, body mass index (BMI) will be calculated, circulating metabolites will be collected, and resting blood pressure will be measured using a standard blood pressure cuff and a stethoscope. The SCAT5 will be conducted by a licensed healthcare professional. For research-specific purposes, body composition will be measured using BIA and C3Logix evaluation will be conducted by trained research personnel. Data collection sheets for the Return-to-Learn Progression, supplement compliance, and GI distress will be collected. If applicable, data collection sheets for the Return-to-Play Progression will be collection. Supplement compliance and GI distress will only be collected at follow up visit #1. Return-to-Learn Progression will be evaluated at each visit until completion of the Return-to-Learn Protocol.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Between the ages of 13 and 19 years
* Acute sports-related concussion

Exclusion Criteria:

* Currently following a low carbohydrate (<100 g/day) diet
* Currently pregnant
* Weight loss greater than or equal to 5% body weight over the last 2 months
* Newly diagnosed and treated (<6 months) mood disorder (i.e. anxiety, depression) or learning disability (i.e. ADD)
* Diagnosed cardiovascular disease, metabolic disease (type 1 or type 2 diabetes), chronic hepatitis, hepatic steatosis, cirrhosis, or IBS
* Presence of a pacemaker, an implanted defibrillator, or other implanted electronic or metallic devices, shrapnel, or other metal
* Previous history of concussion

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 5 (Actual)
Dates: Start 2020-03-20 (Actual); Primary Completion 2022-04-27 (Actual); Study Completion 2022-04-27 (Actual)

PRIMARY OUTCOMES:
Sport Concussion Assessment Tool (SCAT5) | Change in SCAT5 from Baseline to 30 days
  SCAT5 is a standardized tool, not a diagnostic tool, physicians can use for assessing concussions. It will be conducted by a licensed healthcare professional as part of standard of care to obtain numerical values for the following: immediate or on-field assessment (red flags, accident details, etc.), symptom evaluation (dizziness, headache, etc.), cognitive screen (memory, concentration), and neurological screen (balance, coordination). This will be conducted when the concussion occurs and at each clinic visit, irrespective of how much time has passed since the concussion.
C3 Logix System | Change in C3 Logix from Baseline to 30 days
  The computer-based system includes the Graded Symptoms Checklist and Neurological Evaluations. This system is used to assess baseline neurological responses. For assessment, a belt with an iPad holder is affixed to the participant's waist and an iPad is clipped in. Neuro-motor function, balance, and vestibular function are evaluated visual acuity and information processing are assessed. It takes an average of 12 minutes for each athlete to complete the assessment.
Magnetic Resonance Imaging (MRI) | Change in MRI from Baseline to 30 days
  MRI is a noninvasive, routine diagnostic imaging modality that uses a large magnet, radio waves and a computer to produce 2- and 3-dimensional images of the brain. The adolescent will be placed head first into a cylindrical machine that houses a large, tube-shaped magnet that provides a strong magnetic field, so that a radiofrequency coil can image the brain. The magnetic field, along with applied radiofrequency waves, temporarily alters the alignment of hydrogen protons found in water molecules within the body. Computers construct the images based on the radiofrequency signals emitted by the protons.
Serum Analyses | Change in serum levels of glucose and insulin (mg/dL) from Baseline to 14 days to 30 days
  Serum levels of glucose and insulin
Serum Analyses | Change in serum levels of glutamate (µmol/L) from Baseline to 14 days to 30 days
  Serum levels of glutamate
Serum Analyses | Change in serum levels of lactate and ketones (mmol/L) from Baseline to 14 days to 30 days
  Serum levels of lactate and ketones
Serum Analyses | Change in serum levels of TNF, IL-6, and IL-10 (pg/mL) from Baseline to 14 days to 30 days
  Serum levels of TNF, IL-6, and IL-10
Serum Analyses | Change in serum levels of CRP (mg/L) from Baseline to 14 days to 30 days
  Serum levels of CRP

SECONDARY OUTCOMES:
Rate of Completion of Return-to-Learn Protocol | Until completion of the protocol, an average of 3 weeks.
  Progression through the return-to-learn protocol occurs based on the participant's tolerance and will be self-reported. The date each stage is initiated and completed, the total number of days spent in each stage, and the number of attempts needed to complete each stage will be documented on a chart
Rate of Completion of Return-to-Play Protocol | Until completion of the protocol, an average of 3 weeks.
  Progression through the return-to-play protocol will be monitored and documented by athletic trainers at the participant's school once the participant is asymptomatic for at least 48 hours. Initiation and completion dates, number of attempts, symptoms, and post-test Concussion Grading Scales will be recorded by the athletic trainer.
GI Distress Questionnaire | At follow up visit #1 (14 days)
  A questionnaire for five symptoms: nausea, urge to vomit, bloating, belching, and cramps. Participants will be asked to fill out the questionnaire based on their global experience and symptoms throughout the 2-week experimental condition.
Bioelectrical Impedance Analysis (BIA) | The participant will be assessed at baseline (<7 days post-SRC), 14 days, and 30 days
  BIA is a non-invasive technique from which total body composition will be measured. Estimates of fat mass, lean mass, total body water, and bone mineral density for the whole body and defined anatomical region (trunk, arms, and legs) will be assessed using the Tanita body composition analyzer.
Diet Analysis | Immediately after concussion, at first clinic visit (within 7 days after concussion), 14 days after initial visit, 30 days after initial visit, and at each follow up visit up to 1 year
  At each visit participants will be asked to submit a 24-hour dietary recall. A Registered Dietitian will be on site to ensure completeness and clarity. Data from diet recalls will be entered into diet analysis software and examined for total calories, carbohydrate, protein, fat, and select vitamins related to ketone and brain metabolism. Detailed printouts of nutrient intake will be compared to written entries by another member of the research team to identify errors in entry and ensure accurate data entry.
Supplement Compliance | At follow up visit #1 (14 days)
  Throughout the 2-week supplementation period, participants will be asked to verify the supplement is taken 3 times per day.
Anthropometrics | At each visit
  Weight and height (measured with a standard stadiometer with heel plate) will be measured to the nearest 0.1 kilograms and 0.1 inches, respectively, in minimal clothing and without shoes and a z-score for body mass index (BMI) percentiles will be calculated according to age- and sex-standards.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States